CLINICAL TRIAL: NCT04549571
Title: Improving Patient-Centered Communication in Breast Cancer: A RCT of a Shared Decision Engagement System (SHARES)
Brief Title: Improving Patient-Centered Communication in Breast Cancer Through Patient and Provider Interventions
Acronym: SHARES
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Health Services Research
Other Study IDs: A231901CD; NCI-2020-06176 (Registry Identifier: NCI Clinical Trial Reporting Program); UG1CA189823 (NIH); R01CA237046 (NIH)
Record Dates: First submitted 2020-09-09; First posted 2020-09-16 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Anatomic Stage 0 Breast Cancer AJCC v8; Anatomic Stage I Breast Cancer AJCC v8; Anatomic Stage IA Breast Cancer AJCC v8; Anatomic Stage IB Breast Cancer AJCC v8; Anatomic Stage II Breast Cancer AJCC v8; Anatomic Stage IIA Breast Cancer AJCC v8; Anatomic Stage IIB Breast Cancer AJCC v8; Anatomic Stage III Breast Cancer AJCC v8; Anatomic Stage IIIA Breast Cancer AJCC v8; Anatomic Stage IIIB Breast Cancer AJCC v8; Anatomic Stage IIIC Breast Cancer AJCC v8; Prognostic Stage 0 Breast Cancer AJCC v8; Prognostic Stage I Breast Cancer AJCC v8; Prognostic Stage IA Breast Cancer AJCC v8; Prognostic Stage IB Breast Cancer AJCC v8; Prognostic Stage II Breast Cancer AJCC v8; Prognostic Stage IIA Breast Cancer AJCC v8; Prognostic Stage IIB Breast Cancer AJCC v8; Prognostic Stage III Breast Cancer AJCC v8; Prognostic Stage IIIA Breast Cancer AJCC v8; Prognostic Stage IIIB Breast Cancer AJCC v8; Prognostic Stage IIIC Breast Cancer AJCC v8
MeSH Terms: conditions — Breast Carcinoma In Situ | interventions — Interviews as Topic; Practice Guidelines as Topic

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: The enhanced content of the ESE version iCanDecide-ESE is available to the patient, but does not populate differently into the CDB, allowing clinicians to remain blinded to the patient-level randomization arm; therefore, both the patient and the practice and clinicians will be blinded as to which arm the patient is assigned to. However, the surgical practices and their clinicians will know when they are using the CDB so the clinician level intervention will not be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- Arm I: (iCanDecide - ESE) (Experimental): Patients utilize the iCanDecide - ESE website, then undergo surgery within 5 weeks of registration. Patients may also participate in an audio-recorded phone interview over 20 minutes at 9-12 months post registration.
  Interventions: Other: Decision Aid iCanDecide - ESE website; Procedure: Therapeutic Conventional Surgery; Other: Interview; Other: Survey Administration; Other: Quality-of-Life Assessment
- Arm II: (iCanDecide - S) (Active Comparator): Patients utilize the iCanDecide - S website, then undergo surgery within 5 weeks of registration. Patients may also participate in an audio-recorded phone interview over 20 minutes at 9-12 months post registration.
  Interventions: Other: Decision Aid iCanDecide - S website; Procedure: Therapeutic Conventional Surgery; Other: Interview; Other: Survey Administration; Other: Quality-of-Life Assessment
- Clinics 1-5: (CDB) (Experimental): Beginning 4 weeks before the practice begins use of the CDB, clinicians receive training on how to use the CDB and utilize the CDB over weeks 1-60. Clinicians may also participate in an audio-recorded phone interview over 20 minutes.
  Interventions: Other: Interview; Other: Training; Other: Media Intervention; Other: Survey Administration
- Clinics 6-8 (CDB) (Experimental): Beginning 4 weeks before the practice begins use of the CDB, clinicians receive training on how to use the CDB and utilize the CDB over weeks 10-60. Clinicians may also participate in an audio-recorded phone interview over 20 minutes.
  Interventions: Other: Interview; Other: Training; Other: Media Intervention; Other: Survey Administration
- Clinics 9-11 (CDB) (Experimental): Beginning 4 weeks before the practice begins use of the CDB, clinicians receive training on how to use the CDB and utilize the CDB over weeks 20-60. Clinicians may also participate in an audio-recorded phone interview over 20 minutes.
  Interventions: Other: Interview; Other: Training; Other: Media Intervention; Other: Survey Administration
- Clinics 12-14 (CDB) (Experimental): Beginning 4 weeks before the practice begins use of the CDB, clinicians receive training on how to use the CDB and utilize the CDB over weeks 30-60. Clinicians may also participate in an audio-recorded phone interview over 20 minutes.
  Interventions: Other: Interview; Other: Training; Other: Media Intervention; Other: Survey Administration
- Clinics 15-17 (CDB) (Experimental): Beginning 4 weeks before the practice begins use of the CDB, clinicians receive training on how to use the CDB and utilize the CDB over weeks 40-60. Clinicians may also participate in an audio-recorded phone interview over 20 minutes.
  Interventions: Other: Interview; Other: Training; Other: Media Intervention; Other: Survey Administration
- Clinics 18-20 (CDB) (Experimental): Beginning 4 weeks before the practice begins use of the CDB, clinicians receive training on how to use the CDB and utilize the CDB over weeks 50-60. Clinicians may also participate in an audio-recorded phone interview over 20 minutes.
  Interventions: Other: Interview; Other: Training; Other: Media Intervention; Other: Survey Administration
- Clinics 21-25 (usual care) (Active Comparator): Beginning 4 weeks before the practice begins use of the CDB, clinicians receive training on how to use the CDB and continue to provide breast cancer surgical care per their usual care. Clinicians may also participate in an audio-recorded phone interview over 20 minutes.
  Interventions: Other: Interview; Other: Training; Other: Best Practice; Other: Survey Administration

INTERVENTIONS:
Other: Decision Aid iCanDecide - ESE website — Utilize the iCanDecide - ESE website
  Arms: Arm I: (iCanDecide - ESE)
Other: Decision Aid iCanDecide - S website — Utilize the iCanDecide - S website
  Arms: Arm II: (iCanDecide - S)
Procedure: Therapeutic Conventional Surgery — Undergo surgery
  Arms: Arm I: (iCanDecide - ESE); Arm II: (iCanDecide - S)
Other: Interview — Participate in interview
Other: Training — Receive training
  Arms: Clinics 1-5: (CDB); Clinics 12-14 (CDB); Clinics 15-17 (CDB); Clinics 18-20 (CDB); Clinics 21-25 (usual care); Clinics 6-8 (CDB); Clinics 9-11 (CDB)
Other: Media Intervention — Utilize the CDB
  Arms: Clinics 1-5: (CDB); Clinics 12-14 (CDB); Clinics 15-17 (CDB); Clinics 18-20 (CDB); Clinics 6-8 (CDB); Clinics 9-11 (CDB)
Other: Best Practice — Utilize usual care
  Arms: Clinics 21-25 (usual care)
Other: Survey Administration — Ancillary studies
Other: Quality-of-Life Assessment — Ancillary studies
  Arms: Arm I: (iCanDecide - ESE); Arm II: (iCanDecide - S)

SUMMARY:
This trial studies the effectiveness of two interventions on patient reported outcomes of patient centered communication and decision making about breast cancer treatment. The first intervention consists of enhancements to an existing patient-facing breast cancer treatment decision tool called iCanDecide that supports the management of worry, distress, and anxiety as compared to an existing tool. The second intervention consists of a clinician dashboard that populates information after patients view either website regarding any ongoing issues or concerns.

DETAILED DESCRIPTION:
The primary and key secondary objectives of the study:

PRIMARY OBJECTIVES:

I. To demonstrate that the enhanced iCanDecide (iCanDecide-emotional support enhancement [ESE]) intervention is more effective than the standard version (iCanDecide-standard [S]) resulting in higher patient knowledge about locoregional treatment risks and benefits.

II. To demonstrate that the activation of the clinician dashboard (CDB) is more effective than not using a CDB, resulting in higher patient knowledge about locoregional treatment risks and benefits.

SECONDARY OBJECTIVES:

I. To demonstrate that the enhanced iCanDecide (iCanDecide-ESE) intervention is more effective than the standard version (iCanDecide-S), resulting in higher patient-reported breast cancer self-efficacy and lower patient reported cancer worry.

II. To demonstrate that the activation of the clinician dashboard (CDB) is more effective than not using a CDB, resulting in higher patient-reported breast cancer self-efficacy and lower patient reported cancer worry.

OUTLINE: This study is a multi-level trial of SHaDES that has two interventions in a factorial or crossed design: 1) an individually randomized patient-level randomized controlled trial (RCT) to evaluate the standard version (iCanDecide-S) vs. a version with innovative emotional support enhancements (iCanDecide-ESE), and 2) a clinic-level stepped-wedge cluster randomized trial to test a Clinician Dashboard (CDB). Twenty-five surgical practices will be recruited for participation. Practices will be randomized to the timing of the CDB intervention, with some practices initiating the CDB intervention right away, while others may initiate the CDB later or perhaps be randomized to "no CDB" period. Clinicians will be asked to use the CDB beginning in the time period to which their practice was randomized and continuing to the end of the study. After registration, clinicians are followed up at 9 and 18 months. After a patient is registered, the patient will be randomized to one of two arms:

ARM I: Patients utilize the iCanDecide - ESE website, then undergo surgery within 5 weeks of registration. Patients may also participate in an audio-recorded phone interview over 20 minutes at 9-12 months post registration.

ARM II: Patients utilize the iCanDecide - S website, then undergo surgery within 5 weeks of registration. Patients may also participate in an audio-recorded phone interview over 20 minutes at 9-12 months post registration.

After study registration, patients are followed up at 4-5 weeks and 9 months.

Patients will be enrolled at participating clinics during the full duration of the study and all enrolled patients will receive a version of the decision support tool (iCanDecide-S; iCanDecide-ESE). These patient-level activities are not influenced by the timing of the practice-level randomization to the CDB.

ELIGIBILITY:
Inclusion Criteria:

* PATIENT ELIGIBILITY
* Women newly diagnosed with stage 0-III breast cancer. Although men are recommended to undergo surgery to treat breast cancer, male breast cancer is relatively rare and decision making for breast cancer surgery is quite different between men and women
* Planning breast surgery as a component of their definitive treatment within 5 weeks of registration
* Receives care from a clinician and at a practice that has consented to participate in the clinician dashboard practice-level intervention. Practices/clinicians will consent initially at the initiation of the study. Patients will then be identified and recruited in those practices. If a practice has more than one clinician doing breast surgery, patients will be recruited from those clinicians who consent (one or more). Patients of clinicians who have not consented will not be eligible
* Patients must be able to speak English or Spanish with the fluency required to have a direct discussion around treatment decision-making (i.e. without interpreter)
* Age 21-84 years
* CLINICIAN STAKEHOLDER (SURGEONS AND CLINIC STAFF) ELIGIBILITY CRITERIA
* Clinicians eligible for this study include: breast surgeons and their designee(s) (e.g., physician assistants, nurse practitioners, clinical nurse specialists, or nurses) that participate in the treatment decision-making process. At least one surgical oncologist at a practice must agree to participate and sign consent. S/he may then also identify a nurse, physician assistant (PA) or advanced practice provider (APP) with whom s/he works that is involved in the delivery of the care of the same patients to participate. Henceforth, in this protocol they will be referred to as "clinicians"
* Clinicians must agree to have their patients recruited for the entire time the study is open at their practice, which will include time periods in which the clinicians will and time periods in which they will not have access to the CDB
* INSTITUTION ELIGIBILITY:
* Practices that annually provide surgical care for over 100 patients newly diagnosed with breast cancer are eligible to participate in this study
* Eligible practices must have at least one surgical oncologist who agrees to participate in the study

Exclusion Criteria:

* Patients who are visually impaired are not eligible, as they must be able to access the study intervention on a website at home or in clinic and view the decision aid
* Patients with impaired decision-making capacity (such as with a diagnosis of dementia or memory loss) are not eligible for this study
* Practices currently enrolling to Alliance A231701CD are not eligible to participate in this study

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 543 (Actual)
Dates: Start 2021-02-16 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Patient knowledge about risks and benefits of local regional treatment | At 4-5 weeks post patient randomization
  Will be defined as the percentage of correct answers (range: 0-100%) from a 5-item scale previously developed and pilot tested where higher percentages indicate increased knowledge of treatment risks and benefits of local regional treatment. Because the interventions are fully crossed (with intervention and control patients within both intervention and control practices for every time period), the intervention effect of iCanDecide-E and the intervention effect of the clinician dashboard (CDB) will be obtained from a single linear mixed-effects model for the continuous primary outcome measure patient knowledge.

SECONDARY OUTCOMES:
Patient self-efficacy in dealing with breast cancer | At 4-5 weeks post patient randomization
  Will be defined as the composite score obtained from the 11-item (each rated on a 5-point Likert scale: "strongly disagree" to "strongly agree") validated scale designed to assess breast cancer patients' overall feelings of control of their cancer and worry about their cancer (range: 11 to 55); higher scores indicate increased self-efficacy. Because the interventions are fully crossed (with intervention and control patients within both intervention and control practices for every time period), the intervention effect of iCanDecide-E and the intervention effect of the clinician dashboard (CDB) will be obtained from a single linear mixed-effects model for the continuous secondary outcome measure patient self-efficacy.
Patient cancer worry | At 4-5 weeks post patient randomization
  Will be defined as the total score obtained from the 8-item (each rated on a 4-point Likert scale: "never" to "almost always") validated Cancer Worry Scale assessing the degree of cancer-related worry (range: 8 to 40); higher scores indicate more frequent worries about cancer. Because the interventions are fully crossed (with intervention and control patients within both intervention and control practices for every time period), the intervention effect of iCanDecide-E and the intervention effect of the clinician dashboard (CDB) will be obtained from a single linear mixed-effects model for the continuous secondary outcome measure patient cancer worry.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah T. Hawley, PhD, MPH, Study Chair — University of Michigan School of Medicine and Public Health
Locations (27):
- United States (27):
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Helen F Graham Cancer Center, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Kaiser Permanente Moanalua Medical Center, Honolulu, Hawaii
  - SSM Health Good Samaritan, Mount Vernon, Illinois
  - Maine Medical Center- Scarborough Campus, Scarborough, Maine
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Ascension Borgess Hospital, Kalamazoo, Michigan
  - Northern Westchester Hospital, Mount Kisco, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Novant Health Breast Surgery - Greensboro, Greensboro, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - Baptist Memorial Hospital for Women, Memphis, Tennessee
  - ThedaCare Regional Cancer Center, Appleton, Wisconsin
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
  - Ascension Medical Group Southeast Wisconsin - Mayfair Road, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin

REFERENCES:
- [Derived] Hawley ST, Kidwell K, Zahrieh D, McCarthy A, Wills R, Rankin A, Hofer T, Chow S, Jagsi R, Neuman H. Improving patient-centered communication in breast cancer: a study protocol for a multilevel intervention of a shared treatment deliberation system (SharES) within the NCI community oncology research program (NCORP) (Alliance A231901CD). Trials. 2023 Jan 6;24(1):16. doi: 10.1186/s13063-022-07048-4. PMID 36609349